CLINICAL TRIAL: NCT03502876
Title: Tolerance and Resistance to Ibrutinib in Patients With Chronic Lymphocytic Leukemia (CLL): Analysis of Real-life Data: "Snapshot" at 3 Years From the End of Ibrutinib ATU. A National Study of the FILO-LLC Group
Brief Title: Tolerance and Resistance to Ibrutinib in Patients With Chronic Lymphocytic Leukemia (CLL
Status: Completed | Type: Observational
Sponsor: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Other Study IDs: RESISTANCE A L'IBRUTINIB
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: B Cell Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — collection of a blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of the mutational profile of the residual clone and the distribution of lymphocyte subpopulations at 3 years of treatment with ibrutinib

This project has an epidemiological part: to establish the percentage of patients, in a real-life situation, still undergoing treatment 3 years after its initiation, as well as a biological part: to determine the evolution of the clone and the prevalence of BTK mutations and PLCg2 in the absence of clinical or biological criteria for scalability.

DETAILED DESCRIPTION:
Observationnal and biological study

ELIGIBILITY:
Inclusion Criteria:

* patients included in the ATU (epidemiology)
* under treatment at 3 years of ibrutinib
* more than 18 years old

Exclusion Criteria:

* no ibrutinib treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with CLL and treated by ibrutinib in the ATU
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Ibrutinib resistance | under treatment at 3 years of ibrutinib
  In the long term, this study will help to draft new recommendations from FILO-LLC concerning the detection of resistance and the management of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Florence CYMBALISTA, MD PD, Principal Investigator — French Innovative Leukemia Organization
Locations (2):
- France (2):
  - FILO French Innovative Leukemia Organization, Tours
  - Project manager, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FILO internet site — http://www.filo-leucemie.org